CLINICAL TRIAL: NCT01921101
Title: Intensive Nutrition in ARDS: A Clinical Trail (INTACT)
Brief Title: Intensive Nutrition in Acute Respiratory Distress Syndrome (ARDS): A Clinical Trial (INTACT)
Acronym: INTACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: greater mortality in intervention group
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Carol Braunschweig, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 685; NCT01071330 (obsolete NCT alias)
Record Dates: First submitted 2013-07-03; First posted 2013-08-13 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Acute Lung Injury
Keywords: nutrition; enteral feeding; parenteral feeding; hospital malnutrition
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intensive medical nutrition (Other): participants will receive intensive medical nutrition from hospital admission to discharge
  Interventions: Behavioral: intensive medical nutrition
- control (Other): participants will not receive intensive nutritional support from hospital admission to discharge
  Interventions: Other: control

INTERVENTIONS:
Behavioral: intensive medical nutrition — provision of participants energy and protein needs via enteral, parenteral nutrition from hospital admission to discharge
  Arms: intensive medical nutrition
Other: control — participants will receive standard care for nutrition received from hospital admission to discharge
  Arms: control

SUMMARY:
The investigators propose a prospective randomized clinical trail to evaluate the impact of intensive medical nutrition therapy (IMNT) in patients with acute respiratory distress syndrome (ARDS) or acute lung injury (ALI) on short and long-term outcomes. Participant's (N = 200) will be randomized to receive either standard care (SC e.g. ad lib feeding of standard food) or IMNT provided early as enteral nutrition (EN) and continued as intensive diet therapy tailored to maximize oral intake until hospital discharge. Primary outcomes evaluated include infections while hospitalized, immune parameters (CD4 and CD8 cells, serum IL-10 and leptin levels, numbers of T regulatory cells and markers for T cell anergy), days on mechanical ventilation, in the ICU and hospital , and changes in fat free mass(measured by dual energy x-ray absorptiometry), weight, muscular weakness (measured as hand grip strength), fatigue (measured as distanced traveled in 6-minute walk) and pulmonary function.

DETAILED DESCRIPTION:
This study was terminated early due to greater deaths occurring in the intervention group vs the control group. There were a total of 22 deaths, 16 in the intervention and 6 in the control.

ELIGIBILITY:
Inclusion Criteria: Adult patients (> 18 years) with a diagnosis of acute lung injury, with viable GI function for enteral feeding

-

Exclusion Criteria: Patients who are (1) transferred from another ICU, (2) previously admitted to the ICU during the same hospitalization, (3) do not resuscitate status or < 12 month perceived survival due to underlying disease state (4) severely immunosuppressed, (5) immobility prior to ICU admission, (6) documented neurological disease prior to admission. -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: carol l braunschweig, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Sheean PM, Peterson SJ, Chen Y, Liu D, Lateef O, Braunschweig CA. Utilizing multiple methods to classify malnutrition among elderly patients admitted to the medical and surgical intensive care units (ICU). Clin Nutr. 2013 Oct;32(5):752-7. doi: 10.1016/j.clnu.2012.12.012. Epub 2013 Jan 5. PMID 23340043
- [Background] Sheean PM, Peterson SJ, Zhao W, Gurka DP, Braunschweig CA. Intensive medical nutrition therapy: methods to improve nutrition provision in the critical care setting. J Acad Nutr Diet. 2012 Jul;112(7):1073-9. doi: 10.1016/j.jand.2012.02.007. Epub 2012 May 12. PMID 22579721
- [Background] Peterson SJ, Sheean PM, Braunschweig CL. Orally fed patients are at high risk of calorie and protein deficit in the ICU. Curr Opin Clin Nutr Metab Care. 2011 Mar;14(2):182-5. doi: 10.1097/MCO.0b013e3283428e65. PMID 21178611
- [Background] Braunschweig CA, Sheean PM, Peterson SJ. Examining the role of nutrition support and outcomes for hospitalized patients: putting nutrition back in the study design. J Am Diet Assoc. 2010 Nov;110(11):1646-9. doi: 10.1016/j.jada.2010.08.019. PMID 21034876
- [Background] Sheean PM, Peterson SJ, Gurka DP, Braunschweig CA. Nutrition assessment: the reproducibility of subjective global assessment in patients requiring mechanical ventilation. Eur J Clin Nutr. 2010 Nov;64(11):1358-64. doi: 10.1038/ejcn.2010.154. Epub 2010 Aug 11. PMID 20700137
- [Background] Peterson SJ, Tsai AA, Scala CM, Sowa DC, Sheean PM, Braunschweig CL. Adequacy of oral intake in critically ill patients 1 week after extubation. J Am Diet Assoc. 2010 Mar;110(3):427-33. doi: 10.1016/j.jada.2009.11.020. PMID 20184993
- [Result] Braunschweig CA, Sheean PM, Peterson SJ, Gomez Perez S, Freels S, Lateef O, Gurka D, Fantuzzi G. Intensive nutrition in acute lung injury: a clinical trial (INTACT). JPEN J Parenter Enteral Nutr. 2015 Jan;39(1):13-20. doi: 10.1177/0148607114528541. Epub 2014 Apr 9. PMID 24722769
- [Derived] Braunschweig CL, Freels S, Sheean PM, Peterson SJ, Perez SG, McKeever L, Lateef O, Gurka D, Fantuzzi G. Role of timing and dose of energy received in patients with acute lung injury on mortality in the Intensive Nutrition in Acute Lung Injury Trial (INTACT): a post hoc analysis. Am J Clin Nutr. 2017 Feb;105(2):411-416. doi: 10.3945/ajcn.116.140764. Epub 2016 Dec 14. PMID 27974311

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive Medical Nutrition | Control
Started | 40 | 38
Completed | 24 | 32
Not Completed | 16 | 6
Not completed — Death | 16 | 6

BASELINE CHARACTERISTICS:
Population: gender, race/ethnicity, age, diagnosis, admission height and weight, body mass index, ICU admission Acute Physiology and Chronic Health Evaluation II score, Sequential Organ Failure Assessment scores
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Medical Nutrition | Control | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 52.5 (17.1) | 58.6 (16.2) | 55.4 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 19 | 21 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 30 | 27 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 38 | 78
Acute Physiology and Chronic Health Evaluation II (APACHE II) [Mean (Standard Deviation); unit: units on a scale] — The Acute Physiology and Chronic Health Evaluation II (APACHE II) is a severity-of-disease classification. It is applied within 24 hours of admission to the intensive care unit. The scores range from 0-71; higher scores correspond to more severe disease and a higher risk of death
  units on a scale | 23.4 (9.3) | 27.7 (7.9) | 25.5 (8.9)
Sequential Organ Functional Assessment (SOFA) [Mean (Standard Deviation); unit: units on a scale] — The sequential organ failure assessment score (SOFA)is a scoring system used in critically ill patients to assess the extent of their organ function. The total score is based on six different scores, one of the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. These scores range from 0-24; higher scores indicate more severe organ compromise.
  units on a scale | 9.3 (3.8) | 9.4 (3.4) | 9.3 (3.6)
body mass index [Mean (Standard Deviation); unit: Kg/m2] — Body mass index was calculated based on admission weight (Kg)/ height (m)2; NIH classifications for BMI categories were used ( BMI < 18.5 malnourished; 18.5-24.9 normal weight, 25-29.9 overweight and > 30 obese)
  Kg/m2 | 29.8 (9.3) | 30.1 (8.9) | 30 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Infection
Description: All new infections that occurred (including blood, wound, sputum, urinary tract and pulmonary) from enrollment through hospital discharge recorded in the medical record were counted
Time Frame: Assessed daily from study enrollment through hospital discharge, an average of 3 weeks
Measure: Number; unit: participants
Arm/Group | Intensive Medical Nutrition | Control
Number analyzed (Participants) | 40 | 38
participants | 5 | 8
Statistical Analysis 1: Comparison: Intensive Medical Nutrition vs Control; Test type: Superiority or Other; p = 0.29, Chi-squared

2. Secondary Outcome: Length of Hospital Stay
Description: The total number of days the patient is in the hospital
Time Frame: days in hospital
Reporting Status: Not Posted

3. Secondary Outcome: Days on Mechanical Ventilation
Description: the total number of days requiring mechanical ventilation while hospitalized
Time Frame: days
Reporting Status: Not Posted

4. Secondary Outcome: Death
Description: The date of death for all participants that die between enrollment and their final data collection, 24 weeks following hospital discharge
Time Frame: date of occurence
Measure: Number; unit: participants
Arm/Group | Intensive Medical Nutrition | Control
Number analyzed (Participants) | 40 | 38
participants | 16 | 6

5. Other Pre Specified Outcome: Immune Parameters
Description: Markers of immune response (including IL-6, IL-10, adiponectin, leptin, CRP, TNF, CD4/CD8 and HLA/CD14
Time Frame: baseline and weekly while hospitalized
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment throughout hospitalization in all participants, an average of 3 weeks
Description: hyperglycemia, hypoglycemia, aspiration, tube feeding complications, parenteral nutrition complications, death
Arm/Group | Intensive Medical Nutrition | Control
Serious Adverse Events (participants affected / at risk) | 16/40 | 6/38
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Medical Nutrition (N=40) | Control (N=38)
death (General disorders) | 16 (16) | 6 (6) — death from enrollment to 24 weeks post hospital discharge

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No